CLINICAL TRIAL: NCT04231656
Title: Stoke Volume Measurements During Changes in Cardiac Preload: Are Pulse Contour Analysis (CLEARSIGHT) and Transthoracic Bioelectrical Impedance (NICCOMO) Equivalent?
Brief Title: Pulse CONtour and BIoimpedance for Measurements of Stroke Volume During Changes in CARdiac Preload
Acronym: ConBi-Car
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2019_46; 2019-A02697-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Hemodynamic, Monitoring; Anesthesia; Blood Pressure
Keywords: Non-invasive; Stroke volume; Cardiac preload; Interchangeability; Bioelectrical impedance; Pulse contour analysis

STUDY DESIGN:
Intervention Model Description: The primary outcome will be based on measurements performed during a sequence of position changes.
  Sequence A will consist of starting from 0° position, shift to position +20°, then tilt to -20°, and finally back to the 0° position.
  Sequence B will consist of starting from 0° position, shift to position -20°, then tilt to +20°, and finally back to the 0° position.
  Patients will be randomized to take sequence A before the procedure, and then the sequence B at the end of the procedure, or vice-versa (sequence B before sequence A).
  The randomization is not intended to compare the two groups with each other, but only to compensate for a possible"order-effect" in the execution of the maneuvers.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A before sequence B (Experimental): Patients eligible for intermediate risk surgery requiring the placement of an invasive continuous blood pressure measurement device and stroke volume monitoring for fluid management. Sequence A of positioning (before the procedure), and sequence B after the procedure.
  Interventions: Device: CLEARSIGHT and NICCOMO measurements in sequence A; Device: CLEARSIGHT and NICCOMO measurements in sequence B
- Sequence B before sequence A (Experimental): Patients eligible for intermediate risk surgery requiring the placement of an invasive continuous blood pressure measurement device and stroke volume monitoring for fluid management. Sequence B of positioning before the procedure, and sequence A after the procedure.
  Interventions: Device: CLEARSIGHT and NICCOMO measurements in sequence A; Device: CLEARSIGHT and NICCOMO measurements in sequence B

INTERVENTIONS:
Device: CLEARSIGHT and NICCOMO measurements in sequence A — Starting from 0° position, shift to position +20°, then tilt to -20°, and finally back to the 0° position.
  Other Names: CLEARSIGHT and NICCOMO devices (both used during each sequence)
Device: CLEARSIGHT and NICCOMO measurements in sequence B — Starting from 0° position, shift to position -20°, then tilt to +20°, and finally back to the 0° position and collect the last group of figures.
  Other Names: CLEARSIGHT and NICCOMO devices (both used during each sequence)

SUMMARY:
Fluid therapy guided by stroke volume response to repeated fluid challenges is used for hemodynamic optimization during general anesthesia. Two types of devices that measure stroke volume non-invasively are primarily available for intermediate-risk surgery under general anesthesia. They are based on two different techniques, (1) pulse contour analysis, and (2) transthoracic bioimpedance. They have never been compared with each other. Therefore, it is not known (1) whether they are interchangeable for the measurement of stroke volume changes (usually assessed as the "concordance" of two techniques), and (2) whether one is better than the other.

The aim is to study the concordance of these two non-invasive hemodynamic devices. it will use both of them in patients undergoing intermediate risk surgery. They will be tested during modifications of cardiac preload induced by Trendelenburg and anti-Trendelenburg positioning, as well as during intraoperative fluid challenges, vasopressor boluses and alveolar recruitment maneuvers.

DETAILED DESCRIPTION:
The main objective is to assess the concordance of two non-invasive devices using the technology described above : the Clearsight (Edwards Lifesciences, pulse contour analysis), and the Niccomo (Medis, bioimpedance). Both will be used in each patient included in the study. They will be tested during modifications of cardiac preload induced by sequences of position changes (see below) including Trendelenburg and anti-Trendelenburg positioning, performed systematically before and after the procedure, as well as during fluid challenges, vasopressor boluses and alveolar recruitment maneuvers (performed during the procedure according to the needs of the anesthesiologist in charge of the patient). Both monitors will also be compared with an invasive monitor of stroke volume (Vigileo/Flotrac, Edwards Lifesciences), and the respiratory pulse pressure variation will also be measured during the sequences of position changes and will be used as a gold standard for fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Eligible and suitable for intermediate risk surgery, validated by anaesthesia consultation.

There is no definitive definition of intermediate risk. By reference to the literature, surgeries longer than 2 hours (excluding "low risk") and less than 3% postoperative mortality (excluding high-risk surgery). It includes the majority of non-serious visceral (abdominal and gynecological) surgery, plastic or cervical-facial surgery for neoplastic removal or long-term reconstruction, or long-term spinal surgery or neurosurgery of the base of the skull.

- For which the anesthesiologist in charge has planned an invasive monitoring (radial catheter) of arterial blood pressure.

Exclusion Criteria:

* Urgent surgery
* Intracranial hypertension
* Orthostatic hypotension
* Extreme anthropometry: weight >150 kg and 30 kg, size 120 cm and >230 cm
* Related to NICCOMO monitoring:

  * Rhythmic anomaly: Atrial fibrillation, tachycardia with heart rate >200 beats per minute.
  * Aortic disease: Severe sclerosis
  * Valve dysfunction: severe aortic regurgitation,
  * Patient with aortic prosthesis or pacemaker using impedance detection.
  * Occurrence of tachycardia > 200 bpm, occurrence of hypertension with mean arterial pressure >130 mm Hg
  * Simultaneous use of electrical cauterization systems during surgical procedures
  * Septic shock
* Related to CLEARSIGHT monitoring

  * Patient with prior distal perfusion disorders
  * Lower extremity obliterans arteritis stage IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
concordance of stroke volume changes measured with each monitor during the standardized maneuvers of sequences A and B (total: 6 observations per individual). | during each changes of positioning (i.e., for 1-2 minutes in each condition, for a total of 10-15 minutes following initial measurements in basal conditions), during sequences A and B
  4-quadrant plot

SECONDARY OUTCOMES:
Fluid responsiveness defined by areas under the Receiver Operating Characteristic curve (sensitivity and specificity) | during each changes of positioning (i.e., for 1-2 minutes in each condition, for a total of 10-15 minutes following initial measurements in basal conditions), during sequences A and B
  Comparison of areas under the Receiver Operating Characteristic curve (sensitivity and specificity). Each maneuver will be classified as "responder" or "nonresponder" according to the value of Pulse Pressure Variation (PPV) recorded before the maneuver and to the changes in PPV during the maneuver (as previously published)
concordance of stroke volume changes measured with each monitor during the standardized maneuvers mimicking preload decrease. | during each changes of positioning where cardiac preload is supposed to decrease (i.e., for 1-2 minutes in one out of two condition, for a total of 10-15 minutes following initial measurements in basal conditions), during sequences A and B
  4-quadrant plot
concordance of stroke volume changes measured with each monitor during the standardized maneuver mimicking preload increase. | during each changes of positioning where cardiac preload is supposed to increase (i.e., for 1-2 minutes in one out of two condition, for a total of 10-15 minutes following initial measurements in basal conditions), during sequences A and B
  4-quadrant plot
concordance of stroke volume changes measured with each monitor during the surgical procedure (fluid challenges, vasopressor boluses, alveolar recruitment maneuver). | throughout surgery (mean length expected between 3 and 5 hours). Measurements performed during sequences of 5-20 minutes that can occur several times during surgery
  4-quadrant plot
interchangeability of stroke volume measurements with each monitor during sequences A and B | before and after each changes of positioning (i.e., for 1-2 minutes in each condition, for a total of 10-15 minutes following initial measurements in basal conditions), during sequences A and B
  Bland and Altman plot for repeated measures
interchangeability of stroke volume measured with each monitor during the surgical procedure (fluid challenges, vasopressor boluses, alveolar recruitment maneuver). | throughout surgery (mean length expected between 3 and 5 hours). Measurements performed before and after sequences of 5-20 minutes that can occur several times during surgery
  Bland and Altman plot for repeated measures
concordance of stroke volume changes measured with each monitor with that measured by a Vigileo/Flotrac monitor during the standardized maneuvers of sequences A and B (total: 6 observations per individual). | during each changes of positioning (i.e., for 1-2 minutes in each condition, for a total of 10-15 minutes following initial measurements in basal conditions), during sequences A and B
  4-quadrant plot

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Tavernier, MD,PhD, Principal Investigator — University Hospital Lille, France
Locations (1):
- Hôpital Roger Salengro, CHU Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No